CLINICAL TRIAL: NCT02152982
Title: A Phase II/III Randomized Trial of Veliparib or Placebo in Combination With Adjuvant Temozolomide in Newly Diagnosed Glioblastoma With MGMT Promoter Hypermethylation
Brief Title: Temozolomide With or Without Veliparib in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2014-00616; NCI-2014-00616 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A071102; CALGB-A071102; A071102 (Other: Alliance for Clinical Trials in Oncology); A071102 (Other: CTEP); P50CA108961 (NIH); U10CA031946 (NIH); U10CA180821 (NIH)
Record Dates: First submitted 2014-05-27; First posted 2014-06-02 (Estimated); Results first posted 2023-04-04 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Temozolomide; veliparib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (temozolomide, placebo) (Placebo Comparator): Patients receive temozolomide PO QD on days 1-5 and placebo PO BID on days 1-7. Treatment repeats every 28 days for 6 cycles in the absence of disease progression (confirmed progression) or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Other: Quality-of-Life Assessment; Drug: Temozolomide; Drug: Veliparib
- Arm II (temozolomide, veliparib) (Experimental): Patients receive temozolomide as in Arm I and veliparib PO BID on days 1-7. Treatment repeats every 28 days for 6 cycles in the absence of disease progression (confirmed progression) or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Temozolomide; Drug: Veliparib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm I (temozolomide, placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888

SUMMARY:
This randomized phase II/III trial studies how well temozolomide and veliparib work compared to temozolomide alone in treating patients with newly diagnosed glioblastoma multiforme. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether temozolomide is more effective with or without veliparib in treating glioblastoma multiforme.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Test whether the experimental combination of ABT-888 (veliparib) combined with TMZ (temozolomide), compared to the control of placebo combined with TMZ, significantly extends overall survival in newly diagnosed glioblastoma multiforme (GBM) patients with tumor MGMT promoter hypermethylation.

SECONDARY OBJECTIVES:

I. Test whether the experimental treatment significantly extends progression-free survival.

II. Test whether the experimental treatment improves objective tumor response. III. Test whether the experimental treatment is associated with significantly greater rates of grade 3 or higher adverse events.

CORRELATIVE SCIENCE OBJECTIVES:

I. Evaluate the utility of dynamic susceptibility contrast (DSC) and diffusion weighted imaging (DWI) magnetic resonance imaging (MRI) techniques in defining time to progression in the setting of a large multi-institutional clinical trial.

II. Test the concordance between site-determined MGMT methylation status and central laboratory determination of MGMT status in cases with local testing.

III. Evaluate whether genetic or epigenetic alterations in deoxyribonucleic acid (DNA) repair or replication genes are associated with overall survival, progression-free survival, and objective tumor response.

IV. Test whether polymorphisms in MGMT, PARP1, or other DNA repair proteins, are associated with overall survival, progression-free survival, objective tumor response, or rates of grade 3 or higher adverse events.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive temozolomide orally (PO) once daily (QD) on days 1-5 and placebo PO twice daily (BID) on days 1-7. Treatment repeats every 28 days for 6 cycles in the absence of disease progression (confirmed progression) or unacceptable toxicity.

ARM II: Patients receive temozolomide as in Arm I and veliparib PO BID on days 1-7. Treatment repeats every 28 days for 6 cycles in the absence of disease progression (confirmed progression) or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 3 years, every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation: newly diagnosed World Health Organization (WHO) grade IV intracranial glioblastoma or gliosarcoma; GBM with oligodendroglial features are NOT PERMITTED in this study if they are 1p19q codeleted; sites submitting GBM with oligodendroglial features will be asked to provide results of 1p/19q codeletion status
* Sufficient tissue available for central pathology review and MGMT methylation status evaluation
* Patients who have had a local MGMT testing that is unmethylated are not allowed to participate
* Tumor MGMT promoter hypermethylation determined by central testing at MD Anderson
* Confirmation by central pathology review of WHO grade IV glioblastoma or gliosarcoma
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3 (within 14 days prior to study registration)
* Platelets >= 100,000 cells/mm^3 (within 14 days prior to study registration)
* Creatinine =< 1.5 x upper limit of normal (ULN) (within 14 days prior to study registration)
* Bilirubin =< 1.5 x ULN (within 14 days prior to study registration; unless patient has Gilbert's disease)
* Alanine aminotransferase (ALT) =< 3 x ULN (within 14 days prior to study registration)
* Aspartate aminotransferase (AST) =< 3 x ULN (within 14 days prior to study registration)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Measurable disease or non-measurable disease; extent of resection: patients with complete resection, partial resection, or biopsy are eligible
* Progression: patients deemed to have progressive disease based on clinical deterioration after chemoradiation or radiographic progression outside of the radiation field are not eligible; patients deemed to have pseudoprogression are eligible
* Prior treatment:

  * Must have completed standard radiotherapy and concomitant TMZ therapy as defined and determined by the study oncologist
  * Besides concomitant TMZ with radiation, no other therapy (neo-adjuvant or adjuvant) can be given prior to study registration, including chemotherapy (also including Gliadel/carmustine [BCNU] wafers), biologics, immunotherapy, radiation therapy; the only exception is the Optune device (NovoTTF-100A), which may be started any time after end of radiation therapy up through the initiation of Cycle 1; intent to use Optune must be declared at registration for stratification
  * No prior allogeneic bone marrow transplant or double umbilical cord blood transplantation
* Not pregnant and not nursing; females of childbearing potential must have negative urine or serum pregnancy test within 7 days of registration but before start of treatment; a female of childbearing potential is a sexually mature female who:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Concomitant medications: patients receiving anticoagulation should be on stable dose 2 weeks prior to registration
* Comorbid conditions: patients are unable to participate due to the following:

  * Generalized or partial seizure disorder that is uncontrolled at the time of registration; the definition of controlled generalized seizures is patients must be on a stable dose of anti-seizure medication and without generalized seizures for at least 10 days prior to registration; the definition of controlled partial seizures is patients must be on a stable dose of anti-seizure medication for at least 10 days prior to registration; patients with occasional breakthrough partial seizures are allowed at treating physician's discretion
  * Grade 3 or 4 thromboembolic disease within 6 months (mo) of registration
  * Known history of prolonged QT syndrome
* No history of major surgery =< 14 days prior to registration
* Patients must have adequate organ and marrow function measured within 28 days prior to administration of ABT-888 as defined below:

  * >= 10.0 g/dL hemoglobin (Hb) with no blood transfusion in the past 28 days
* No Patients with treatment-related acute myeloid leukemia (AML) (t-AML)/myelodysplastic syndrome (MDS) or with features suggestive of AML/MDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2025-12-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jann N Sarkaria, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (392):
- United States (391):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - John Muir Medical Center-Concord, Concord, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - The NeuroMedical Center-Clinic, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - New England Cancer Specialists - Topsham, Topsham, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - John F Kennedy Medical Center, Edison, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - East Carolina University, Greenville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Fundacion De Investigacion de Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Sarkaria JN, Ballman KV, Kizilbash SH, Sulman EP, Giannini C, Friday BB, Butowski NA, Mohile NA, Piccioni DE, Battiste JD, Drappatz J, Campian JL, Mashru S, Jaeckle KA, O'Brien BJ, Dixon JG, Kabat BF, Laack NL, Hu LS, Kaufmann T, Kumthekar P, Ellingson BM, Anderson SK, Galanis E. Efficacy of Adding Veliparib to Temozolomide for Patients With MGMT-Methylated Glioblastoma: A Randomized Clinical Trial. JAMA Oncol. 2024 Dec 1;10(12):1637-1644. doi: 10.1001/jamaoncol.2024.4361. PMID 39480453
- [Derived] Gupta SK, Kizilbash SH, Carlson BL, Mladek AC, Boakye-Agyeman F, Bakken KK, Pokorny JL, Schroeder MA, Decker PA, Cen L, Eckel-Passow JE, Sarkar G, Ballman KV, Reid JM, Jenkins RB, Verhaak RG, Sulman EP, Kitange GJ, Sarkaria JN. Delineation of MGMT Hypermethylation as a Biomarker for Veliparib-Mediated Temozolomide-Sensitizing Therapy of Glioblastoma. J Natl Cancer Inst. 2015 Nov 27;108(5):djv369. doi: 10.1093/jnci/djv369. Print 2016 May. PMID 26615020

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Temozolomide, Placebo): Patients receive temozolomide as in Arm II and placebo PO BID on days 1-7. Treatment repeats every 28 days for 6 cycles in the absence of disease progression (confirmed progression) or unacceptable toxicity. > > Laboratory Biomarker Analysis: Correlative studies >
  * Placebo Administration: Given PO >
  * Quality-of-Life Assessment: Ancillary studies >
  * Temozolomide: Given PO
- Arm II (Temozolomide, Veliparib): Patients receive temozolomide PO QD on days 1-5 and veliparib PO BID on days 1-7. Treatment repeats every 28 days for 6 cycles in the absence of disease progression (confirmed progression) or unacceptable toxicity. > > Laboratory Biomarker Analysis: Correlative studies >
  * Quality-of-Life Assessment: Ancillary studies >
  * Temozolomide: Given PO >
  * Veliparib: Given PO
Period: Overall Study
Arm/Group | Arm I (Temozolomide, Placebo) | Arm II (Temozolomide, Veliparib)
Started | 224 | 223
Started Treatment | 213 | 218
Completed | 144 | 134
Not Completed | 80 | 89
Not completed — Withdrawal by Subject | 17 | 16
Not completed — Did not start treatment | 11 | 5
Not completed — Disease progression | 41 | 52
Not completed — Adverse Event | 7 | 12
Not completed — Complicating disease | 1 | 1
Not completed — Death | 0 | 3
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Temozolomide, Placebo): Patients receive temozolomide as in Arm II and placebo PO BID on days 1-7. Treatment repeats every 28 days for 6 cycles in the absence of disease progression (confirmed progression) or unacceptable toxicity. > > Laboratory Biomarker Analysis: Correlative studies >> Placebo Administration: Given PO >> Quality-of-Life Assessment: Ancillary studies >> Temozolomide: Given PO
- Arm II (Temozolomide, Veliparib): Patients receive temozolomide PO QD on days 1-5 and veliparib PO BID on days 1-7. Treatment repeats every 28 days for 6 cycles in the absence of disease progression (confirmed progression) or unacceptable toxicity. > > Laboratory Biomarker Analysis: Correlative studies >> Quality-of-Life Assessment: Ancillary studies >> Temozolomide: Given PO >> Veliparib: Given PO
- Total: Total of all reporting groups
Arm/Group | Arm I (Temozolomide, Placebo) | Arm II (Temozolomide, Veliparib) | Total
Number analyzed (Participants) | 224 | 223 | 447
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (12.40) | 58.8 (11.55) | 58.5 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 96 | 190
  Male | 130 | 127 | 257
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 208 | 212 | 420
  Unknown or Not Reported | 7 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 6 | 17
  White | 197 | 199 | 396
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 14 | 25
Extent of Resection [Count of Participants; unit: Participants] — How much of the glioblastoma was removed with surgery; gross total resection is associated with more positive disease outcomes than subtotal resection or biopsy.
  Participants
    Gross total resection | 140 | 140 | 280
    Subtotal resection or biopsy | 84 | 83 | 167
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG performance status quantifies how able a patient is to care for themselves and continue regular activity. The scale ranges from 0 (fully active, no restrictions due to disease) to 5 (dead).
  Participants
    0-1 | 205 | 205 | 410
    2 | 19 | 18 | 37
Side of Lesion [Count of Participants; unit: Participants]
  Bilateral | 3 | 8 | 11
  Left | 107 | 106 | 213
  Midline | 1 | 2 | 3
  Right | 113 | 107 | 220
Tumor Location [Count of Participants; unit: Participants]
  Multiple locations | 82 | 74 | 156
  Frontal | 67 | 65 | 132
  Occipital | 3 | 9 | 12
  Other | 1 | 3 | 4
  Parietal | 26 | 24 | 50
  Temporal | 42 | 45 | 87
  Thalamus | 3 | 3 | 6
Planned concomitant use of Optune device [Count of Participants; unit: Participants] — Patients had the option to continue using a NovoTTF-100A (Optune) device during treatment
  Participants
    No | 191 | 194 | 385
    Yes | 33 | 29 | 62

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The distribution of OS for each arm will be estimated using the Kaplan-Meier method and compared with a stratified logrank test.
Time Frame: 83 months
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Arm I (Temozolomide, Placebo): Patients receive temozolomide as in Arm II and placebo PO BID on days 1-7. Treatment repeats every 28 days for 6 cycles in the absence of disease progression (confirmed progression) or unacceptable toxicity. > > Laboratory Biomarker Analysis: Correlative studies >
  > Placebo Administration: Given PO >
  > Quality-of-Life Assessment: Ancillary studies >
  > Temozolomide: Given PO
- Arm II (Temozolomide, Veliparib): Patients receive temozolomide PO QD on days 1-5 and veliparib PO BID on days 1-7. Treatment repeats every 28 days for 6 cycles in the absence of disease progression (confirmed progression) or unacceptable toxicity. > > Laboratory Biomarker Analysis: Correlative studies >
  > Quality-of-Life Assessment: Ancillary studies >
  > Temozolomide: Given PO >
  > Veliparib: Given PO
Arm/Group | Arm I (Temozolomide, Placebo) | Arm II (Temozolomide, Veliparib)
Number analyzed (Participants) | 224 | 223
months | 24.8 [22.6 to 27.7] | 28.1 [24.3 to 33.3]
Statistical Analysis 1: Comparison: Arm I (Temozolomide, Placebo) vs Arm II (Temozolomide, Veliparib); Test type: Superiority; p = 0.1673, Log Rank

2. Secondary Outcome: Interaction With Optune Device
Description: Cox proportional hazards model will be used to evaluate whether there is a potential interaction between the treatment arm and the Optune device. If an interaction is detected, separate analyses of treatment effect (using Cox models) will be done for patients treated with the Optune device and patients who were not treated with the Optune device.
Time Frame: 10 years
Population: Analysis population is patients that reported actual optune use
Measure: Number; unit: participants
Arm/Group | Arm I (Temozolomide, Placebo) | Arm II (Temozolomide, Veliparib)
Number analyzed (Participants) | 224 | 223
participants
  Reporting actual Optune use | 42 | 42
  No actual Optune use | 182 | 181
Statistical Analysis 1: Comparison: Arm I (Temozolomide, Placebo) vs Arm II (Temozolomide, Veliparib); Test type: Other — Interaction test; p = 0.6659, Type 3 likelihood-ratio p-value; Cox Proportional Hazard = 0.89, 95% CI 2-sided [0.53 to 1.50]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: The distribution of PFS for each arm will be estimated using the Kaplan-Meier method, and be compared using Cox proportional hazard models with all stratification factors adjusted. Progression (PD): Defined by any of the following:
  1. > 25% increase in sum of products of perpendicular diameters of enhancing lesions, compared with the smallest tumor measurement obtained either at baseline or best response
  2. Significant increase in T2/FLAIR non-enhancing lesion on stable or increasing doses of corticosteroids compared with baseline scan or best response after therapy initiation (stable doses of steroids include patient not on steroids) not caused by comorbid events
  3. Any new lesion
  4. Clear clinical deterioration not attributable to other causes apart from tumor or change in corticosteroid dose
  5. Failure to return for evaluation as a result of death or deteriorating condition
  6. Clear progression of non-measurable disease
Time Frame: 120 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Temozolomide, Placebo) | Arm II (Temozolomide, Veliparib)
Number analyzed (Participants) | 224 | 223
months | 12.1 [10.6 to 14.9] | 13.2 [10.5 to 14.9]
Statistical Analysis 1: Comparison: Arm I (Temozolomide, Placebo) vs Arm II (Temozolomide, Veliparib); Test type: Superiority; p = 0.3164, Stratified Log Rank; Stratified Cox Proportional Hazard = 1.05, 95% CI 2-sided [0.86 to 1.29]

4. Secondary Outcome: Objective Tumor Response
Description: Defined as complete response (CR) or partial response (PR) as specified in the Revised Assessment in Neuro-Oncology (RANO) criteria. An objective tumor response will be evaluated for each patient and the tumor response count will be summarized for each arm and compared using the Chi-square test. For CR, all of the following must be true:
  disappearance of all enhancing measurable and non-measurable disease; no new enhancing lesions; stable or improved non-enhancing lesions; patients must be off corticosteroids; stable or improved clinically A PR requires all of the following: > 50% decrease in sum of products of perpendicular diameters of all measurable enhancing lesions compared with baseline; no progression of non-measurable disease; no new lesions; stable or improved non-enhancing lesions on same or lower dose of corticosteroids compared with baseline scan; steroid dose should be same or lower compared with baseline scan; stable or improved clinically
Time Frame: 5 years
Population: All patients randomized to the trial with measurable disease per RANO criteria at registration and at one or more assessment(s) post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Temozolomide, Placebo) | Arm II (Temozolomide, Veliparib)
Number analyzed (Participants) | 118 | 119
Participants | 34 | 37
Statistical Analysis 1: Comparison: Arm I (Temozolomide, Placebo) vs Arm II (Temozolomide, Veliparib); Test type: Superiority; p = 0.7018, Chi-squared

5. Secondary Outcome: Overall Adverse Event Rates for Grade 3 or Higher Adverse Events
Description: Assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (version 5 beginning April 1, 2018). The overall adverse event rates for grade 3 or higher adverse events will be summarized and be compared using Chi-Square or Fisher's Exact tests between treatment arms. The maximum grade for each type of treatment-related adverse event will be recorded for each patient, and frequency tables for each arm will be reviewed to determine patterns. Treatment-related adverse events will be tabulated for each arm.
Time Frame: 5 years
Population: Only includes patients that began treatment
Measure: Number; unit: participants with at least 1 grade 3+ AE
Arm/Group | Arm I (Temozolomide, Placebo) | Arm II (Temozolomide, Veliparib)
Number analyzed (Participants) | 213 | 218
participants with at least 1 grade 3+ AE | 93 | 133
Statistical Analysis 1: Comparison: Arm I (Temozolomide, Placebo) vs Arm II (Temozolomide, Veliparib); Test type: Superiority; p = 0.0003, Chi-squared

6. Other Pre Specified Outcome: Change in Quality of Life (QOL)
Description: Measured by the fatigue/uniscale tool. The fatigue/uniscale tool will be used as a measure of QOL. Potential differences in fatigue levels of patients treated on the two different arms will be evaluated. Changes in this measure will be evaluated over the course of treatment for both arms and will be compared using a two-sample t-test at each timepoint. Will also compute a normalized area under the curve (AUC) for the values of each patient over time and compare the mean AUCs for patients on the two arms.
Time Frame: Baseline to up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: MGMT Status
Description: The concordance between site-determined MGMT methylation status and central laboratory determination of MGMT status will be analyzed using the Chi-Square test of proportions and 95% confidence intervals for the proportion of tests in disagreement with the local site.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality monitored/assessed for up to 83 months; Adverse Events monitored/assessed for up to 5 years
Arm/Group | Arm I (Temozolomide, Placebo) | Arm II (Temozolomide, Veliparib)
All-Cause Mortality (participants affected / at risk) | 175/213 | 183/218
Serious Adverse Events (participants affected / at risk) | 47/213 | 43/218
Other Adverse Events (participants affected / at risk) | 207/213 | 217/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Temozolomide, Placebo) (N=213) | Arm II (Temozolomide, Veliparib) (N=218)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (6) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (11) | 7 (7)
Fever (General disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 5 (6)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Edema cerebral (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 2 (2)
Muscle weakness right-sided (Nervous system disorders) | 0 (0) | 2 (2)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 5 (5) | 7 (7)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 3 (3)
Confusion (Psychiatric disorders) | 4 (7) | 3 (4)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (2)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (8) | 1 (4)
Thromboembolic event (Vascular disorders) | 4 (4) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Temozolomide, Placebo) (N=213) | Arm II (Temozolomide, Veliparib) (N=218)
Anemia (Blood and lymphatic system disorders) | 17 (36) | 36 (84)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 0 (0) | 3 (4)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 6 (11) | 3 (3)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 2 (5)
Flashing lights (Eye disorders) | 1 (1) | 0 (0)
Periorbital edema (Eye disorders) | 1 (2) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (3)
Constipation (Gastrointestinal disorders) | 99 (294) | 94 (256)
Diarrhea (Gastrointestinal disorders) | 40 (85) | 45 (88)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 2 (7)
Dysphagia (Gastrointestinal disorders) | 2 (4) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (7) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 129 (367) | 126 (355)
Vomiting (Gastrointestinal disorders) | 15 (18) | 19 (29)
Chills (General disorders) | 4 (5) | 2 (3)
Death NOS (General disorders) | 1 (1) | 2 (2)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 3 (5) | 3 (5)
Fatigue (General disorders) | 182 (744) | 181 (734)
Fever (General disorders) | 4 (5) | 0 (0)
Gait disturbance (General disorders) | 2 (10) | 4 (4)
Gen disord and admin site conds-Oth spec (General disorders) | 3 (4) | 4 (4)
Neck edema (General disorders) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 2 (2)
Allergic reaction (Immune system disorders) | 2 (4) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (2)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 2 (4)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 2 (3) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 1 (2)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (5) | 6 (11)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Fracture (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (8) | 12 (20)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (5) | 5 (8)
Blood bilirubin increased (Investigations) | 1 (3) | 3 (8)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 2 (2)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 3 (6) | 3 (4)
Investigations - Other, specify (Investigations) | 1 (5) | 2 (7)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 60 (186) | 60 (177)
Neutrophil count decreased (Investigations) | 45 (93) | 115 (282)
Platelet count decreased (Investigations) | 116 (382) | 191 (667)
Weight gain (Investigations) | 2 (2) | 3 (8)
Weight loss (Investigations) | 9 (23) | 8 (22)
White blood cell decreased (Investigations) | 27 (61) | 62 (170)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 88 (244) | 83 (207)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (24) | 16 (21)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 4 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (4) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4) | 7 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (13) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (10) | 8 (16)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (6) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (7)
Amnesia (Nervous system disorders) | 1 (4) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 2 (8)
Cognitive disturbance (Nervous system disorders) | 4 (4) | 4 (5)
Concentration impairment (Nervous system disorders) | 2 (7) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 9 (26) | 12 (20)
Dysarthria (Nervous system disorders) | 2 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (5) | 7 (18)
Dysphasia (Nervous system disorders) | 2 (6) | 3 (3)
Edema cerebral (Nervous system disorders) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 109 (328) | 99 (284)
Hydrocephalus (Nervous system disorders) | 1 (1) | 2 (2)
Lethargy (Nervous system disorders) | 2 (3) | 3 (3)
Memory impairment (Nervous system disorders) | 6 (13) | 10 (26)
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 1 (2)
Muscle weakness right-sided (Nervous system disorders) | 0 (0) | 5 (6)
Nervous system disorders - Oth spec (Nervous system disorders) | 2 (18) | 3 (23)
Paresthesia (Nervous system disorders) | 2 (2) | 3 (8)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (6) | 0 (0)
Seizure (Nervous system disorders) | 27 (44) | 30 (57)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 2 (7) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (7)
Confusion (Psychiatric disorders) | 4 (6) | 4 (8)
Depression (Psychiatric disorders) | 3 (6) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (6) | 2 (2)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 3 (7)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 1 (2) | 2 (4)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 4 (4)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Testicular disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 8 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (6) | 8 (11)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (7)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 1 (2)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 7 (16) | 6 (15)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 4 (10) | 2 (2)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT02152982/Prot_SAP_000.pdf